CLINICAL TRIAL: NCT05930002
Title: Role of Ivermectin and Colchicine in Treatment of COVID-19: Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, hemat abdelsalam ahmed, Assistant lecturer of family medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Drugs in COVID-19
Record Dates: First submitted 2023-06-22; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: Ivermectin; Colchecine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Colchicine

STUDY DESIGN:
Intervention Model Description: Three arm randomized controlled clinical trial
Who Masked: Participant
Masking Description: Using sealed envelopes for either participants or controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ivermectin group (Active Comparator): received standard treatment plus Ivermectin in the form of oral tablets (0.2 mg/kg/day) single dose on an empty stomach for three successive days
  Interventions: Drug: Ivermectin Tablets
- Colchicine group (Active Comparator): received standard treatment plus Colchicine 0.5mg tablets (3times/day after meal for 3 days then twice daily for 4 days)
  Interventions: Drug: Colchicine 0.5 MG
- Control group (Active Comparator): received the standard treatment according to the protocol of the Egyptian Supreme Council of University Hospitals (http://scu.eg/pages/university_hospitals) (Vitamin C 500mg tablet twice daily, Vitamin D3 2000-4000 IU/day, Zinc 75mg tablet once daily for two weeks and needed protocol of management according to case assessment and severity)
  Interventions: Drug: Standared managment

INTERVENTIONS:
Drug: Ivermectin Tablets — oral tablets (0.2 mg/kg/day) single dose on an empty stomach for three successive days.
  Other Names: Iverzine
  Arms: Ivermectin group
Drug: Colchicine 0.5 MG — 0.5mg tablets (3times/day after meal for 3 days then twice daily for 4 days)
  Other Names: Colchicine
  Arms: Colchicine group
Drug: Standared managment — (Vitamin C 500mg tablet twice daily, Vitamin D3 2000-4000 IU/day, Zinc 75mg tablet once daily for two weeks
  Arms: Control group

SUMMARY:
Corona virus disease 2019 (COVID-19) is caused by severe acute respiratory syndrome corona virus 2 (SARS-CoV-2), a new corona virus that emerged in Wuhan, China, in December 2019. It spread rapidly throughout the world causing great mortality. Till date, there is no specific treatment for COVID-19; Ivermectin and colchicine were proposed as therapeutic options for treatment of COVID-19. Our randomised controlled clinical trial aims to assess the effectiveness of ivermectin and colchicine for treating COVID-19.

DETAILED DESCRIPTION:
Patients will be selected from Triage/COVID-19 Outpatient Clinic and every patients will be subjected to the following:

1. Clinical history will be obtained about socio-demographic data such as age, gender, residence, marital status, smoking history...etc, medical history including (weight, current medication, symptoms (onset, course, duration) and presence of Co-morbidities.
2. Full general examination including: temperature, heart rate, blood pressure, respiratory rate and oxygen saturation.

   Suspected patients according to CDC criteria will be subjected to laboratory and radiological confirmation with (PCR-COVID-19, Complete Blood Count, CRP, Ferritin and D-Dimer) and High resolution CT chest.

   After confirmation of the diagnosis and patients are classified as moderate with laboratory and radiological findings.

   o Grouping: All patients enrolled in the study according the calculated sample size will be equally divided randomly into 3 groups using sealed envelope contain code for each group.
   * Group A (Ivermectin group): COVID-19 patients with moderate severity who will receive standard treatment according to the protocol of the Egyptian Supreme Council of University Hospitals plus Ivermectin in the form of oral tablets e.g. (Iverzine 6mg) (200 mcg/kg/day) (4 tablets in the first day and then 2 tablet in the second and third day) on an empty stomach (Kaur et al., 2021).

   Iverzine:

   • Manufactured by: Unipharma Pharmaceutical Chemicals Co.

   • Side effects of iverzine: Abdominal pain, Asthenia, Hypotension and Headache (Fujimoto et al., 2014).

   o Group B (Colchicine group): COVID-19 patients with moderate severity who will receive standard treatment according to the protocol of the Egyptian Supreme Council of University Hospitals plus Colchicine 0.5mg tablets (3times/day after meal for 3 days then twice daily for 4 days) (Karatza et al., 2021).

   Then all groups will receive instructions of home isolation.

   Colchicine:

   • Manufactured by: El Nasr Pharmaceutical Chemicals Co.

   • Side effects of Colchicine: Gastro intestinal side effects e.g abdominal pain, vomiting, diarrhoea (Imazio et al., 2014).

   o Group C (Control group): COVID-19 patients with moderate severity who will receive standard treatment according to the protocol of the Egyptian Supreme Council of University Hospitals (still not published) (Vitamin C 500mg tablet twice daily, Vitamin D3 2000-4000 IU/day, Zinc 75mg tablet once daily for two weeks and needed protocol of management according to case assessment and severity).

   o Randomization: The researcher will use sealed envelopes containing code for intervention or control.

   o Follow up: Participants will be followed up twice weekly by telephone evaluating their symptoms (increase or decrease, duration of symptoms and development of new symptoms) compliance on treatment, daily measurement of temperature, oxygen saturation, need for oxygen inhalation, need for hospital admission, ICU admission, mechanical ventilation, mortality and improvement of inflammatory markers (CBC, CRP, Ferritin and D-dimer).

   o Final evaluation: Discharge from isolation after 10 days after symptom onset or10 days after their first positive swab (Teranaka et al., 2021).

   Participants will be asked about improvement of symptoms or residual symptoms. Inflammatory markers (CBC, CRP, Ferritin and D-dimer) will be re-tested on day 14 then after 1 month from onset of symptoms.

   o End point: The study will be continued up to complete the sample size, improvement of patient's symptoms, no development of new symptoms, need for hospitalization or ICU admission and Occurrence of adverse events (AES) or serious adverse events (SAEs) throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged (18-64) years with confirmed criteria of COVID-19 infection.
* Moderate Cases: Patients have symptoms (such as fever, respiratory tract symptoms), pneumonic manifestations can be seen in chest imaging and oxygen saturation more than 94% (Egyptian Ministry of Health and Population, 2020).

Exclusion Criteria:

* Pregnant or lactating female.
* Any co-morbidities (DM, hypertension, Asthma……etc.).
* Participants receiving immunosuppressive or chemotherapy drugs.
* Active malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
duration and number of symptoms | one month
  Participants were followed up twice weekly for one month. They were called by phone to ask about their symptoms e.g: they were asked about symptoms relief, number of symptoms, duration of symptoms e.g cough, fever (temperature measurement by thermometer)
Concentration of inflammatory markers (CBC, CRP, Ferritin and D-dimer ) | one month
  Patients were asked to do inflammatory markers (CBC, CRP, Ferritin and D-dimer ) in the first 5 days as initial labs .
  Two weeks later, patients were followed up in the clinic. They were asked to repeat the primary investigations (CBC, CRP, Ferritin and D-dimer).
  After one month of symptoms onset, patients were followed up in the clinic and the previous investigations (CBC, CRP, Ferritin and D-dimer) were re-tested
need for oxygen inhalation | one month
  Patients were asked to measure oxygen saturation daily and according to the measurement, the need for oxygen was determined.
need for hospital admission, ICU admission, mechanical ventilation and mortality. | one month
  Patients were assessed for the need of hospital admission, ICU admission, mechanical ventilation or if mortality documented. all these measures were done according to oxygen saturation measurement , investigations and assessment of symptoms if they improve or deteriorate

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No